CLINICAL TRIAL: NCT02499276
Title: Comparative Effects of Variable Pressure Support, Neurally Adjusted Ventilatory Assist (NAVA) and Proportional Assist Ventilation (PAV) on the Variability of the Breathing Pattern and on Patient Ventilator Interaction
Brief Title: Comparative Effects of Variable Pressure Support, NAVA and PAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADOREPS-2013-0802
Record Dates: First submitted 2015-06-12; First posted 2015-07-16 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-07

CONDITIONS: Respiratory Failure
Keywords: mechanical ventilation; pressure support ventilation; NAVA; PAV; variable ventilation; patient ventilator asynchrony
MeSH Terms: conditions — Respiratory Insufficiency; Patient-Ventilator Asynchrony

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PSV, PAV, NAVA, Variable-PSV (Experimental): This is a crossover study in which each patient will be ventilated in the following modes of mechanical ventilation: Pressure Support Ventilation (PSV), Neurally Adjusted Ventilator Assist (NAVA), Proportional assist ventilation (NAVA) and variable Pressure Support Ventilation (Variable-PSV), in a randomised order.
  Interventions: Device: PSV, NAVA, PAV, Variable-PSV

INTERVENTIONS:
Device: PSV, NAVA, PAV, Variable-PSV — Each patient enrolled in the study will be ventilated in all the following modes: PSV, NAVA, PAV and variable PSV

SUMMARY:
Experimental animal data suggest that increasing breathing pattern variability in mechanical ventilation could be beneficial. Variable ventilation can be induced through the following modes: Neurally Adjust Ventilatory Assist (NAVA), Proportional Assist Ventilation (PAV) and Variable-Pressure Support Ventilation (V-PSV). These modes have not yet been compared to each other. Pilot observations in our department suggest a feasibility in patients.

The objectives of the study are to compare the impact of PSV, NAVA, PAV and V-PSV on the variability of the breathing pattern, patient-ventilator asynchrony, risk of lung overdistension, gas exchange, and repartition of ventilation.

DETAILED DESCRIPTION:
Cross-over, prospective, randomized controlled monocentric trial . Patients on pressure support ventilation will be ventilated with PSV, NAVA, PAV, and V-PSV (in a randomized sequence).

In each mode the level of assistance will be set to achieve a similar tidal volume of 6-8 ml/kg.

The following data will be measured and recorded: airway flow and pressure, electrical activity of the diaphragm (EAdi), blood gases, electrical impedance tomography, end tidal partial pressure in carbon dioxide (PEtCO2).

Will be calculated: the coefficient of variation (CV, standard deviation (SD)/mean) of the peak pressure (Ppeak), EAdi and of the main descriptors of the breathing pattern, the prevalence of the main patient-ventilator asynchronies, the prevalence of tidal volume (VT) >10ml/kg, ventrodorsal repartition of ventilation and inhomogeneity index, dead space

ELIGIBILITY:
Inclusion Criteria:

* patient on mechanical ventilation for >48 h
* estimated duration of mechanical ventilation >24h
* hemodynamic stability

Exclusion Criteria:

* pregnancy
* impossibility to insert an EAdi catheter
* neuromuscular disease, phrenic nerve lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation of the tidal volume (VT) | 1 hour
  Coefficient of variation (standard deviation/mean) of the tidal volume (VT)
Coefficient of variation of the respiratory rate (RR) | 1 hour
  Coefficient of variation (standard deviation/mean) of the respiratory rate (RR)
Coefficient of variation of the inspiratory time (Ti) | 1 hour
  Coefficient of variation (standard deviation/mean) of the inspiratory time (Ti)
Coefficient of variation of the electrical activity of the diaphragm (EAdi) | 1 hour
  Coefficient of variation (standard deviation/mean) of the electrical activity of the diaphragm (EAdi)
Coefficient of variation of the maximal inspiratory pressure (Ppeak) | 1 hour
  Coefficient of variation (standard deviation/mean) of the maximal inspiratory pressure (Ppeak)

SECONDARY OUTCOMES:
Patient ventilator asynchrony | 1 hour
  asynchrony index (composite outcome, that includes double triggering, auto triggering and ineffective efforts) )
Safety from lung overdistension, assessed by the proportion of tidal volumes (VT) >10 ml/kg | 1 hour
Gas exchanges | 6 hours
  Ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2), arterial carbon dioxide pressure (PaCO2)
Repartition of ventilation measured by electrical impedance tomography | 6 hours
Dead space to tidal volume ratio (Vd/Vt) | 6 hours
  Vd/Vd, is a ratio between two volumes

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Demoule, MD, PHD, Study Director — Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil
Locations (1):
- Service de Pneumologie et Réanimation Médicale, Groupe Hospitalier Pitié Salpêtrière, Paris, France